CLINICAL TRIAL: NCT06868706
Title: Virtual Reality-Supported Video Modeling for Enhancing Motor Skill Acquisition in Swimming
Brief Title: VR-Based Video Modeling for Novice Swimmers
Acronym: VR-Swim Skill
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Erzurum Technical University (Other)
Collaborators: Ataturk University (Other)
Responsible Party: Principal Investigator, Deniz Bedir, Associate Professor Doctor, Erzurum Technical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: ETU-VR-2025-02; E-70400699-000-2100187704 (Other: Ataturk University)
Record Dates: First submitted 2025-02-27; First posted 2025-03-11 (Actual); Last update posted 2025-03-11 (Actual); Status verified 2025-03

CONDITIONS: Skills Acquisition; Sports Performance; Swimming
Keywords: Virtual reality; Video modeling; Swimming performance; Motor skill acquisition; Novice swimmers

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- VR-Supported Video Modeling Group (Experimental): Participants receive traditional swimming training as well as VR-supported video modelling training.
  Interventions: Behavioral: VR-Supported Video Modeling; Behavioral: Traditional Swimming Training
- Traditional Swimming Group (Active Comparator): Participants only receive traditional swimming training, but no VR or video modelling.
  Interventions: Behavioral: Traditional Swimming Training

INTERVENTIONS:
Behavioral: VR-Supported Video Modeling — Participants receive virtual reality (VR) supported video modeling training in addition to traditional swimming training.
  Arms: VR-Supported Video Modeling Group
Behavioral: Traditional Swimming Training — Participants receive only traditional swimming training. Individuals in this group learn swimming techniques through traditional methods (practising in the water under the supervision of an instructor).

SUMMARY:
Understanding the complex dynamics of motor skill acquisition in swimming is critical for developing effective training programs. Advances in technology, such as virtual and augmented reality, offer new opportunities to enhance learning and performance in this field. This study investigated the impact of virtual reality (VR)-supported video modeling (VM) swimming exercise programs compared with traditional approaches on the swimming performance of beginners.

Fifty-five university students participated in the study. They were divided into two groups: the VR-supported VM group (VRVM) (n=28) and the traditional swimming group (TSG) (n=27). The VRVM group engaged in VR-supported VM practice in addition to traditional swimming training, whereas the TSG group only participated in traditional swimming training. The performance variables measured included swimming stroke (SS), crawling kick (CK), swimming duration (SD), heart rate (HR), and rate of perceived excretion (RPE).

ELIGIBILITY:
Inclusion Criteria:

Never having taken a swimming course before. Not having any health problems. Not having water phobia.

Exclusion Criteria:

To be able to progress by stroking on the water without any support from anywhere.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2023-02-27 (Actual); Primary Completion 2023-06-02 (Actual); Study Completion 2023-10-17 (Actual)

PRIMARY OUTCOMES:
Swimming stroke | Post-Intervention (After 11 Weeks)
  Swimming stroke (SS) refers to the number of strokes performed per minute, which impacts a swimmer's propulsion through the water. It is a critical factor in determining speed and efficiency.
Swimming duration | Post-Intervention (After 11 Weeks)
  The swimming duration is the swimmer's time to cover a 25-meter distance. Swimmers using the proper freestyle technique are expected to cover a given distance in less time, with lower SD scores positively contributing to swimming performance.
Crawling kick | Post-Intervention (After 11 Weeks)
  The crawling kick plays an essential role in a swimmer's propulsion and overall speed and balance in the water. Novice swimmers may focus more on breathing and arm strokes, neglecting foot strokes (Lucero, 2015). Therefore, this study assumes that more foot strokes positively impact performance. The CK was calculated based on the number of foot strokes performed over a 25-meter distance.

SECONDARY OUTCOMES:
Heart rate | Post-Intervention (After 11 Weeks)
  Heart rate is the parameter used to monitor the physiological response of swimmers to exercise and to assess aerobic fitness.

CONTACTS AND LOCATIONS:
Locations (1):
- Erzurum Technical University Faculty of Sport Sciences, Erzurum, Yakutiye, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Franklin ZC, Wright DJ, Holmes PS. Using Action-congruent Language Facilitates the Motor Response during Action Observation: A Combined Transcranial Magnetic Stimulation and Eye-tracking Study. J Cogn Neurosci. 2020 Apr;32(4):634-645. doi: 10.1162/jocn_a_01510. Epub 2019 Dec 10. PMID 31820678
- [Background] Craig AB Jr, Pendergast DR. Relationships of stroke rate, distance per stroke, and velocity in competitive swimming. Med Sci Sports. 1979 Fall;11(3):278-83. PMID 522640
- [Background] Clark SE, Ste-Marie DM. The impact of self-as-a-model interventions on children's self-regulation of learning and swimming performance. J Sports Sci. 2007 Mar;25(5):577-86. doi: 10.1080/02640410600947090. PMID 17365543
- [Background] Calvo-Merino B, Glaser DE, Grezes J, Passingham RE, Haggard P. Action observation and acquired motor skills: an FMRI study with expert dancers. Cereb Cortex. 2005 Aug;15(8):1243-9. doi: 10.1093/cercor/bhi007. Epub 2004 Dec 22. PMID 15616133
- [Background] Barbosa TM, Bragada JA, Reis VM, Marinho DA, Carvalho C, Silva AJ. Energetics and biomechanics as determining factors of swimming performance: updating the state of the art. J Sci Med Sport. 2010 Mar;13(2):262-9. doi: 10.1016/j.jsams.2009.01.003. Epub 2009 May 5. PMID 19409842
- [Background] Araiza-Alba, P., Keane, T., Matthews, B., Simpson, K., Strugnell, G., Chen, W. S., & Kaufman, J. The potential of 360-degree virtual reality videos to teach water-safety skills to children, Computers & Education, 2021, 163.